CLINICAL TRIAL: NCT04972955
Title: Predicting Dysglycemia in Individuals With Gestational Diabetes Immediately Postpartum Using Continuous Glucose Monitoring
Acronym: PREDISPOSE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Jennifer Yamamoto, MD, University of Manitoba
Other Study IDs: REB20-1660
Record Dates: First submitted 2021-06-28; First posted 2021-07-22 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes; Prediabetes; Complicating Pregnancy; Type 2 Diabetes; Pregnancy Related; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases
Keywords: Gestational Diabetes; Pregnancy; Prediabetes; Prospective Cohort Study; Type 2 Diabetes; CGM; Continuous Glucose Monitoring; Flash Glucose Monitoring; Screening
MeSH Terms: conditions — Diabetes, Gestational; Prediabetic State; Pregnancy Complications; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women diagnosed with gestational diabetes: Pregnant individuals who have been diagnosed with gestational diabetes during the current pregnancy
  Interventions: Device: Freestyle Libre 2

INTERVENTIONS:
Device: Freestyle Libre 2 — Participants will wear a continuous glucose monitoring device, the Freestyle Libre 2, for two weeks following delivery.
Device: Freestyle Libre 2 — Participants will wear a second continuous glucose monitoring device, the Freestyle Libre 2, for two weeks at 4-6 months postpartum and before their standard of care postpartum bloodwork after having gestational diabetes.

SUMMARY:
Gestational diabetes is one of the most common medical disorders in pregnancy and is a major risk factor for the postpartum development of dysglycemia. Despite the high risk of developing dysglycemia, 50-80% of women with gestational diabetes are not receiving testing within a year postpartum. The investigators will conduct a prospective cohort study to examine the use of continuous glucose monitoring immediately postpartum to estimate the risk of maternal dysglycemia postpartum.

DETAILED DESCRIPTION:
Gestational diabetes is one of the most common medical disorders in pregnancy and affects up to 18% of pregnancies. It is associated with an increased risk of both maternal and neonatal complications. Importantly, gestational diabetes is a major risk factor for the postpartum development of pre-diabetes or type 2 diabetes (together referred to as dysglycemia). Specifically, half of people with gestational diabetes will develop dysglycemia within 10 years of delivery. Despite the high risk of developing dysglycemia, 50-80% of women with recent gestational diabetes are not receiving testing within a year postpartum.

There are likely many factors contributing to this low screening rate. These include individual factors such as socioeconomic status and maternal age, as well as the nature of the guideline recommended test itself. The Diabetes Canada 2018 Clinical Practice Guidelines recommend screening for maternal dysglycemia between "6 weeks to 6 months postpartum" with a 75g oral glucose tolerance test (OGTT). This recommendation is based on expert opinion. While the 75g OGTT is thought to be the "gold-standard" for screening for dysglycemia postpartum, it has many pitfalls. First, the OGTT is widely disliked by women as it is time consuming and inconvenient. It requires consuming a sugary drink in addition to two separate venipunctures. Second, the 75g OGTT is notoriously unreproducible. Finally, it takes only a "snap shot" of a woman's glucose and insulin response with only two measurements over two-hours.

Emerging technologies are changing the landscape of diabetes care. Continuous glucose monitoring (Freestyle Libre 2) is one such technology. People easily insert a small cannula just under the skin using an applicator. While the device is in place, it measures interstitial glucose concentrations every 15 minutes. It is a small disc (~size of a quarter) and it can be worn during typical daily activities such as sleeping, showering, and exercising. The sensor can store up to 8 hours of glucose readings in 15-minute intervals. People scan the sensor using a smartphone or reader to upload glucose readings to the Freestyle Libre 2 app, which can be viewed by a clinician and/or researcher. Continuous glucose monitoring gives a detailed picture of glycemic excursions throughout the day including both fasting and postprandial states.

There are currently no published studies examining the use of continuous glucose monitoring postpartum. Furthermore, no studies have examined continuous glucose monitoring's potential role in diagnosis of maternal dysglycemia postpartum. There is an unmet need to improve postpartum screening for individuals with gestational diabetes so that high risk individuals do not miss the opportunity for early treatment. To address this, the investigators will perform a study examining the use of continuous glucose monitoring immediately postpartum to estimate the risk of maternal dysglycemia postpartum. This is an observational study which aims to see if CGM can be used to diagnose diabetes. The CGM device in this study will be used for diagnosis and not as an intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals age 18 and older
* Diagnosed with gestational diabetes by the Diabetes Canada guidelines (including both the preferred or alternate testing approaches) or have an HbA1c of 6.0-6.4% during pregnancy
* Have any of the following: have an elevated fasting glucose (≥ 5.3 mmol/L) on the diagnostic 75g OGTT in pregnancy; required insulin or metformin for treatment during pregnancy; body mass index (BMI) ≥ 25kg/m^2, yes/no (<27 weeks gestation BMI of ≥25 kg/m^2 or ≥27 weeks gestation predicted BMI of ≥ 25 kg/m^2 using (current weight in kg - 10kg)/height in meters^2)
* Planned in-hospital delivery
* Able to provide informed consent
* Willingness to use the study device and complete assessments postpartum
* Have access to email in order to complete participant questionnaire through REDCap

Exclusion Criteria:

* A clinical diagnosis of non-gestational diabetes (i.e., pre-existing type 1 or 2 diabetes) prior to or during pregnancy
* Planned x-ray, MRI or CT within 3 weeks postpartum
* Has an implantable medical device (ex. pacemaker)
* On medications known to affect glucose metabolism (for example glucocorticoids, metformin etc.) while wearing the CGM postpartum
* On medications which may interfere with the Freestyle Libre 2 accuracy (for example Vitamin C >1000mg/day) while wearing the CGM postpartum
* Unable to speak and understand French or English
* Unable to consent or declined informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who are currently pregnant and have been diagnosed with gestational diabetes during the current pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of CGM as a screening test for postpartum dysglycemia. | 1-14 days postpartum; 4-6 months postpartum
  Diagnostic accuracy will be measured as sensitivity, specificity, positive likelihood ratio and negative likelihood ratio.

SECONDARY OUTCOMES:
New diagnosis of maternal diabetes or prediabetes based on HbA1c alone, and a combination of the 75-gram OGTT and the HbA1c. | 4-6 months postpartum
  Diabetes or prediabetes based on the postpartum 75-gram OGTT will be evaluated as fasting plasma glucose ≥7.0 mmol/L or 2-hour plasma glucose of ≥11.1 mmol/L or fasting plasma glucose 6.1-6.9 mmol/L or 2-hour plasma glucose of 7.8-11.1 mmol/L, respectively. Diabetes or prediabetes based on the postpartum HbA1c will be evaluated as ≥6.5 and ≥6.0%, respectively. Diabetes and prediabetes will be analyzed separately and together.
Acceptability of CGM based on an acceptability questionnaires after device return and after final testing. | 15-17 days postpartum; 4-6 months postpartum
  The Acceptability Questionnaires for the Freestyle Libre 2 Postpartum will be completed at two points throughout the study. "Strongly agree/painless" and "agree/almost painless" will be considered as "rated favorably" in planned analyses.
Dyslipidemia at time of postpartum bloodwork. | 4-6 months postpartum
  Dyslipidemia is defined as abnormal levels of lipids in the bloodstream, which elevate cardiovascular risk. Lactation state will be recorded given impacts on lipid levels.
Glycemic variability reflected by coefficients of variation and standard deviations of blood glucose data. | 1-14 days postpartum; 4-6 months postpartum
  Blood glucose data will be collected using the Freestyle Libre 2 continuous glucose monitoring system.
Cardiometabolic and related health outcomes diagnosed by regular healthcare team. | 1, 2 and 5 years postpartum
  Information on dysglycemia, hypertension, cardiovascular disease, and additional health outcomes will be obtained through administrative provincial databases and chart review.
Cost component analysis of CGM vs. 75g OGTT. | 4-6 months to 5 years postpartum
  Costs of assessing blood glucose via CGM versus lab-derived OGTT results will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Yamamoto, MD, Principal Investigator — University of Manitoba
Locations (4):
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Mount Sinai Hospital, Toronto, Ontario
  - Universite Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Sellers EA, Dean HJ, Shafer LA, Martens PJ, Phillips-Beck W, Heaman M, Prior HJ, Dart AB, McGavock J, Morris M, Torshizi AA, Ludwig S, Shen GX. Exposure to Gestational Diabetes Mellitus: Impact on the Development of Early-Onset Type 2 Diabetes in Canadian First Nations and Non-First Nations Offspring. Diabetes Care. 2016 Dec;39(12):2240-2246. doi: 10.2337/dc16-1148. Epub 2016 Oct 4. PMID 27703026
- [Background] Lowe WL Jr, Scholtens DM, Lowe LP, Kuang A, Nodzenski M, Talbot O, Catalano PM, Linder B, Brickman WJ, Clayton P, Deerochanawong C, Hamilton J, Josefson JL, Lashley M, Lawrence JM, Lebenthal Y, Ma R, Maresh M, McCance D, Tam WH, Sacks DA, Dyer AR, Metzger BE; HAPO Follow-up Study Cooperative Research Group. Association of Gestational Diabetes With Maternal Disorders of Glucose Metabolism and Childhood Adiposity. JAMA. 2018 Sep 11;320(10):1005-1016. doi: 10.1001/jama.2018.11628. PMID 30208453
- [Background] Ferrara A, Peng T, Kim C. Trends in postpartum diabetes screening and subsequent diabetes and impaired fasting glucose among women with histories of gestational diabetes mellitus: A report from the Translating Research Into Action for Diabetes (TRIAD) Study. Diabetes Care. 2009 Feb;32(2):269-74. doi: 10.2337/dc08-1184. Epub 2008 Nov 4. PMID 18984776
- [Background] McGovern A, Butler L, Jones S, van Vlymen J, Sadek K, Munro N, Carr H, de Lusignan S. Diabetes screening after gestational diabetes in England: a quantitative retrospective cohort study. Br J Gen Pract. 2014 Jan;64(618):e17-23. doi: 10.3399/bjgp14X676410. PMID 24567578
- [Background] Butalia S, Donovan L, Savu A, Johnson J, Edwards A, Kaul P. Postpartum Diabetes Testing Rates after Gestational Diabetes Mellitus in Canadian Women: A Population-Based Study. Can J Diabetes. 2017 Dec;41(6):613-620. doi: 10.1016/j.jcjd.2016.12.013. Epub 2017 May 12. PMID 28506815
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Feig DS, Berger H, Donovan L, Godbout A, Kader T, Keely E, Sanghera R. Diabetes and Pregnancy. Can J Diabetes. 2018 Apr;42 Suppl 1:S255-S282. doi: 10.1016/j.jcjd.2017.10.038. No abstract available. PMID 29650105
- [Background] Neiger R, Coustan DR. The role of repeat glucose tolerance tests in the diagnosis of gestational diabetes. Am J Obstet Gynecol. 1991 Oct;165(4 Pt 1):787-90. doi: 10.1016/0002-9378(91)90418-q. PMID 1951534
- [Background] Meltzer SJ, Snyder J, Penrod JR, Nudi M, Morin L. Gestational diabetes mellitus screening and diagnosis: a prospective randomised controlled trial comparing costs of one-step and two-step methods. BJOG. 2010 Mar;117(4):407-15. doi: 10.1111/j.1471-0528.2009.02475.x. Epub 2010 Jan 26. PMID 20105163
- [Derived] Sigurdson SM, Bernier KJ, Donovan LE, Feig DS, Lemieux P, Pylypjuk C, Shen GX, Jiang D, Nerenberg K, Chrisp MM, Katz PM, Benham JL, Yamamoto JM. Predicting dysglycaemia in individuals with gestational diabetes immediately postpartum using continuous glucose monitoring (PREDISPOSE) in a multicentre prospective cohort study in Canada: a study protocol. BMJ Open. 2025 Jul 30;15(7):e103771. doi: 10.1136/bmjopen-2025-103771. PMID 40738649